CLINICAL TRIAL: NCT05892900
Title: Transcutaneous Vagus Nerve Stimulation (tVNS) to Acutely Reduce Emotional Vulnerability and Improve Emotional Regulation in Borderline Personality Disorder (tVNS-BPD): a Randomized, Single-blind, Sham-controlled Trial
Brief Title: Transcutaneous Vagus Nerve Stimulation (tVNS) for Borderline Personality Disorder (tVNS-BPD)
Acronym: tVNS-BPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Giuseppe Guerriero, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tVNS-BPD-001; SU-971761 (Other Grant/Funding Number: Sahlgrenska University Hospital); CIVID:22-10-041068 (Registry Identifier: Swedish Medical Products Agency (Läkemedelsverket))
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Borderline Personality Disorder
Keywords: transcutaneous vagus nerve stimulation; borderline personality disorder; emotional vulnerability; emotion regulation
MeSH Terms: conditions — Borderline Personality Disorder; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous vagus nerve stimulation (tVNS) (Experimental): 1 tVNS session of ca 45 minutes
  The electrodes are placed at the left ear concha. The ear concha is principally innerved by the afferent branch of the vagus nerve
  Interventions: Device: Transcutaneous vagus nerve stimulation (tVNS)
- Sham Transcutaneous vagus nerve stimulation (tVNS) (Sham Comparator): 1 sham tVNS session of ca 45 minutes
  The electrodes are attached to the center of the left ear lobe, which is known to be free of cutaneous vagal innervation
  Interventions: Device: Sham transcutaneous vagus nerve stimulation (Sham tVNS)

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation (tVNS) — The electrodes are placed at the left ear concha. The ear concha is principally innerved by the afferent branch of the vagus nerve
  Other Names: Transcutaneous auricular vagus nerve stimulation (taVNS)
  Arms: Transcutaneous vagus nerve stimulation (tVNS)
Device: Sham transcutaneous vagus nerve stimulation (Sham tVNS) — The electrodes are attached to the center of the left ear lobe, which is known to be free of cutaneous vagal innervation
  Other Names: Sham Transcutaneous auricular vagus nerve stimulation (Sham taVNS)
  Arms: Sham Transcutaneous vagus nerve stimulation (tVNS)

SUMMARY:
The goal of this clinical trial is to test the efficacy of transcutaneous vagus nerve stimulation (tVNS) in borderline personality disorder. The main question it aims to answer is:

• Is tVNS effective in acutely reducing emotional reactivity in borderline personality disorder?

Participants will be randomized to a single session of tVNS or sham-tVNS while going through an affect-inducing procedure. It will consist of the presentation of one neutral and three negative affect-inducing videos in sequence, each of which is followed by a post-induction period during which participants will rate the quality and intensity of their current self-reported emotions.

Researchers will compare the tVNS and sham tVNS groups to see if there is a difference in the intensity of the self-reported emotions between the groups.

DETAILED DESCRIPTION:
The study will be a randomized, single-blind, sham-controlled trial. The goal of this clinical trial is to test the efficacy of transcutaneous vagus nerve stimulation (tVNS) acutely reduce emotional vulnerability and improve emotional regulation in borderline personality disorder. The main questions it aims to answer are:

* Is tVNS effective in acutely reducing emotional reactivity in borderline personality disorder?
* Is tVNS effective in acutely reducing baseline emotional arousal in borderline personality disorder?
* Is tVNS effective in acutely ease emotional recovery in borderline personality disorder?
* Is tVNS effective in acutely improve emotional regulation in borderline personality disorder?

The participants will be randomized to a single session of tVNS or sham-tVNS while going through an affect induction procedure. It will consist of the presentation of one neutral and three negative affect-evoking 4-minutes-long videos in sequence, each of which is followed by a 4-minutes post-induction period during which participants will rate the quality and intensity of their current self-reported emotions (post-induction ratings) and the perceived effectiveness in managing their emotions during the video presentation. The rating of the current self-reported emotions will be repeated after every post-induction period (recovery ratings).

To test the difference in negative emotional arousal at every stage and the perceived effectiveness in managing emotions between the tVNS and sham tVNS groups, mixed models with individuals as random effects will be used. These models will take into account the repeated measurements of the same individuals at baseline, pre-induction, post-induction, and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Swedish-speaking and able to provide informed consent to participate in the study
* Female and between the ages 18 and 50 years old.
* Current DSM-5 (Diagnostic and statistical manual of mental disorder-5) diagnosis of BPD based on the Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD)
* Capable (in the Investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Any unstable medical and/or neurological condition
* Currently pregnant
* Any significant neurological disorder or condition likely to be associated with increased intracranial pressure or cognitive impairment (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis)
* Current diagnosis of delirium, dementia or another cognitive disorder secondary to a general medical condition
* Established diagnosis of a developmental and neuropsychiatric disorder (e.g. Down syndrome, autism-spectrum disorder, ADHD)
* Non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the affect induction procedure, follow and answer the survey instructions and questions)
* Alcohol or substance use disorder (relating to opioids, cocaine, amphetamine or benzodiazepine) currently or within the past 1 month
* Daily treatment with antiepileptics (e.g., carbamazepine, gabapentin, lamotrigine, levetiracetam, pregabalin, sodium valproate, topiramate) or benzodiazepines (last dose over 7 days before the screening)
* Alcohol or substance use disorder (relating to opioids or cocaine) currently or within the past 1 month
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* History or diagnosis of bipolar or chronic psychotic disorder (e.g., schizophrenia, schizoaffective disorder).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in negative emotional arousal from baseline at immediately after affect-induction (post-induction ratings) as assessed by PANAS | Baseline and immediately after every of the four videos.
  The emotional arousal will be measured through the self-reported ratings of negative emotions on the PANAS (PANAS-N). The scale uses adjectives that describe mood states rather than discrete emotions and are rated from 1 = very slightly or not at all to 5 = extremely.

SECONDARY OUTCOMES:
Change in negative emotional arousal from baseline at prior to affect-induction (pre-induction ratings) as assessed by PANAS | Baseline and 4 minutes after the tVNS/sham tVNS has begun, before the affect induction procedure.
  The emotional arousal will be measured through the self-reported ratings of negative emotions on the PANAS (PANAS-N). The scale uses adjectives that describe mood states rather than discrete emotions and are rated from 1 = very slightly or not at all to 5 = extremely.
Change in negative emotional arousal from immediately after affect-induction at 4 minutes after affect induction (recovery ratings) as assessed by PANAS | Immediately after and at 4 minutes after every of the three affect inducing videos
  The emotional arousal will be measured through the self-reported ratings of negative emotions on the PANAS (PANAS-N). The scale uses adjectives that describe mood states rather than discrete emotions and are rated from 1 = very slightly or not at all to 5 = extremely.
Perceived effectiveness in managing emotions (PEME) during affect induction. | Immediately after every of the four videos
  Participants will be asked during the post-induction period about their perceived effectiveness in managing their emotions (PEME) by asking them to rate "How difficult was it to manage your emotional response to this film clip?" from 1 = not at all to 9 = extremely. This scale will be interpreted as a subjective difficulty in regulating emotions in response to each video stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Steinn Steingrimsson, MD, PhD, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Giuseppe Guerriero, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
This will be discussed if the occasion arises in order to follow GDPR rules

REFERENCES:
- [Background] Daros AR, Williams GE, Jung S, Turabi M, Uliaszek AA, Ruocco AC. More is not always better: Strategies to regulate negative mood induction in women with borderline personality disorder and depressive and anxiety disorders. Personal Disord. 2018 Nov;9(6):530-542. doi: 10.1037/per0000296. Epub 2018 Jul 12. PMID 29999393
- [Background] Guerriero G, Wartenberg C, Bernhardsson S, Gunnarsson S, Ioannou M, Liljedahl SI, et al. Efficacy of transcutaneous vagus nerve stimulation as treatment for depression: A systematic review. J Affect Disord Rep. 2021 Dec 1;6:100233. https://doi.org/10.1016/j.jadr.2021.100233
- [Derived] Guerriero G, Liljedahl SI, Carlsen HK, Lopez Munoz M, Daros AR, Ruocco AC, Steingrimsson S. Transcutaneous auricular vagus nerve stimulation to acutely reduce emotional vulnerability and improve emotional regulation in borderline personality disorder (tVNS-BPD): study protocol for a randomized, single-blind, sham-controlled trial. Trials. 2024 Jun 19;25(1):397. doi: 10.1186/s13063-024-08230-6. PMID 38898522